CLINICAL TRIAL: NCT07304193
Title: Clinical and Genetic Aspects of Fetuses With Sex-chromosome Disorders
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 1-10-72-170-23
Record Dates: First submitted 2025-12-12; First posted 2025-12-26 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Sex Chromosome Disorders
Keywords: Turner syndrome; Klinefelter syndrome; XYY syndrome; XXX syndrome
MeSH Terms: conditions — Sex Chromosome Disorders; Turner Syndrome; Klinefelter Syndrome; 47, XYY syndrome; Triple X syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Fetal tissue and placental tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Electively aborted fetuses with genetically verified sex chromosome abnormalities
- Elective aborted health fetuses

SUMMARY:
To conduct a comprehensive clinical investigation of electively aborted fetuses with sex chromosome disorders and their placentas, in parallel with analyses of epigenetic alterations and changes in gene expression in these fetuses and their placentas, with the aims to:

1. delineate how variations in sex chromosome number affect the epigenetic and genetic mechanisms regulating gene expression in the placenta and in multiple fetal tissues in fetuses with sex chromosome disorders;
2. identify the epigenetic and genetic mechanisms and placental and fetal alterations that underlie the phenotypic manifestations observed in fetuses with sex chromosome disorders.

ELIGIBILITY:
Inclusion criteria cases:

* Age ≥18 years
* Fetuses with genetically verified sex chromosome disorders
* Gestational age between 11+0 and 22+6 at the time of abortion or at delivery due to intrauterine fetal death
* Written informed consent

Inclusion criteria cases:

* Age ≥18 years
* No known sex chromosome disorder or other genetic disorder in the fetus
* No known fetal malformations
* Fetal growth within the normal range
* Gestational age between 11+0 and 22+6 at the time of abortion

Ages: 11 Weeks to 22 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Recruitent of cases will take place at obstetric departments and departments of clinical genetics throughout Denmark.
  Recruitment of controls will take place at obstetric departments in the Central Denmark Region.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
DNA methylation profile | 5 years
  DNA methylation of placenta DNA methylation across fetal tissues
Gene expression profile | 5 years
  RNA expression of placenta RNA expression across fetal tissue

CONTACTS AND LOCATIONS:
Overall Officials: Anne Skakkebæk, MD, PHD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark